CLINICAL TRIAL: NCT07040774
Title: Natural History of Type 1 Interferonopathies: Insights From a European Cohort
Acronym: EU-IFNp
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HJ-24- EU-IFNp
Record Dates: First submitted 2025-06-12; First posted 2025-06-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Genetic Disease; Immune Dysfunction; Neurological Diseases or Conditions; Autoimmune Diseases
Keywords: Immune dysfuntion; Neurological disease; Autoimmune diseases; Genetics diseases; Interferon; Aicardi-Goutieres Syndrom
MeSH Terms: conditions — Genetic Diseases, Inborn; Immune System Diseases; Autoimmune Diseases; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with genetically confirmed type I interferonopathy

SUMMARY:
Type I interferonopathies are rare autoinflammatory disorders caused by genetic defects and associated with significant morbidity and mortality. These diseases are refractory to conventional immunosuppressive therapies. They typically occur in childhood, although disease onset in adulthood has been observed. The clinical spectrum is wide and mainly involves the central nervous system. Joint involvement is also common, and more rarely, haematological features such as cytopenias or immunodeficiency may be observed.

Nearly all patients show consistent over-activation of the type I IFN pathway, as evidenced, the expression of IFN-stimulated genes, the so-called 'interferon signature'. To date, the natural history of interferonopathies remains unclear.

In this context, the establishment of a natural history of type I interferonopathy in patients is proposed to elucidate the pathophysiological mechanisms and identify biomarkers for diagnosis, prognosis, and disease activity, with the aim of better characterising the diversity of interferonopathies.

The main objective is to characterise the evolution of the pathology in paediatric and adult patients with type I interferonopathies.

The overall aim of this research is to propose therapeutic options tailored to patient phenotypes and to better define patient sub-groups in order to optimise the preparation of future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed patient with type I interferonopathy
* Patient affiliated to a social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

- Opposition of the patient and/or parental authority if the patient is a minor, to participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with genetically confirmed type I interferonopathy in Europe. 500 patients estimated.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2045-05 (Estimated); Study Completion 2045-05 (Estimated)

PRIMARY OUTCOMES:
Characterizing disease progression in pediatric and adult patients with type I interferonopathies | 2025-2045
  Composite description of phenotypes of patients with type I interferonopathies according to genotype (clinical, biological) over time.

SECONDARY OUTCOMES:
Identifing and characterising genotype-specific immunological factors | 2025-2045
  Description of specific immunological factors according to genotype
Research of biomarkers for diagnosis, prognosis and monitoring of disease activity | 2025-2045
  Biomarkers identified for diagnosis, prognosis and monitoring of disease activity
Monitoring of treatment response according to phenotype and genotype | 2025-2045
  Treatment response by phenotype and genotype

CONTACTS AND LOCATIONS:
Locations (32):
- Medical University Innsbruck, Innsbruck, Austria
- Antwerp University Hospital, Antwerp, Belgium
- Children's Hospital Zagreb, Zagreb, Croatia
- Motol University Hospital, Prague, Czechia
- France (21):
  - CHU d'Angers, Angers
  - Hôpital de Mercy - CHR Metz Thionville, Ars-Laquenexy
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU Morvan, Brest
  - Hôpital Femme Mère Enfant - HCL, Bron
  - CHU de Dijon, Dijon
  - Hôpitaux Nord Ouest Villefranche, Gleizé
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Claude Huriez, CHU de Lille, Lille
  - APHM Hôpitaux de Marseille, Marseille
  - CHU de Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU de Nantes, Nantes
  - CH Agen-Nérac, Nérac
  - Hôpital de l'Archet, Nice
  - Hôpital Armand Trousseau, Paris
  - Hôpital Bichat, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital des Enfants - CHU de Toulouse, Toulouse
  - Hôpital Necker Enfants Malades, Paris, Île-de-France Region
- University of Tübingen, Tübingen, Germany
- Meyer Children's Hospital IRCCS, Florence, Italy
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Son Espases, Palma de Mallorca
- Karolinska University Hospital, Stockholm, Sweden
- Hacettepe İhsan Doğramacı Children's Hospital, Ankara, Turkey (Türkiye)
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom